CLINICAL TRIAL: NCT05748509
Title: COMPARISON OF THE LUMBAR EXTANSOR MUSCLES' ACTIVATIONS DURING DIFFERENT LOW BACK EXERCISES
Brief Title: COMPARISON OF THE LUMBAR EXTANSOR MUSCLES' ACTIVATIONS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-141
Record Dates: First submitted 2023-02-20; First posted 2023-02-28 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Low Back Pain
Keywords: Lumbal Lordosis; Thoracic Kyphosis; Muscle Activation; Low Back Exercises
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Surface EMG activations — We will try to find out which of the exercises such as pressing the back back, waist extension on the balance ball, lumbar extension in the active prone position, Superman exercises have better lumbar extensor muscle activations. Muscle activations of individuals will be evaluated using superficial EMG. An 8-channel EMG Noraxon MiniDTS system (Noraxon, USA, Inc, Scottsdale, AZ) will be used to measure signals from the muscles.

SUMMARY:
Low back pain is a public health problem faced by 65-80% of the world's population at some point in their lives. Although the prognosis for low back pain is considered good, 80% of patients with acute low back pain recover within 6 weeks, and 7-10% of them have complaints that last longer than 3 months and become chronic, causing great labor and economic loss.

A multidisciplinary approach is often required in the treatment of low back pain, which is one of the most common diseases in the society and one of the most expensive diseases in terms of both labor loss and treatment cost. In this approach, waist exercises and waist protection training are accepted as an effective and economical method. In our society, there is no conscious education and exercise habits about the techniques of protecting back health. Most patients with chronic low back pain initially ignore low back pain, but apply to health centers when symptoms related to low back pathology become severe. In many studies, it has been shown that strong waist and abdominal muscles and good physical condition reduce musculoskeletal damage in low back traumas. Most studies show that back extensors and flexors are of low strength in patients with low back pain compared to asymptomatic individuals. In the study conducted by Lee et al. on 3000 male workers, it was found that low back pain was lower in those with exercise habits. In a systematic review and meta-analysis conducted in 2017, it was reported that leisure time physical activity can reduce the risk of chronicity of nonspecific low back pain by 11-16%.

When the literature is examined, it is seen that there are different exercise approaches recommended for the conservative treatment of low back pain. There are studies reporting that pilates is effective in terms of pain, disability, kinesiophobia, function, quality of life, flexibility and balance in patients with low back pain and that it has no harmful effects. In another study, it was reported that traditional Chinese exercises are effective in terms of pain, disability and cognitive function in low back pain, and interventions performed 1-2 times a week and 3-4 times a week are associated with reduced pain. Liu et al. In a study conducted in 2019 by Chen-style Tai Chi in individuals aged 50 years and older with chronic nonspecific low back pain, it was found that Chen style Tai Chi reduced pain but did not improve lower extremity proprioception. Wieland et al. showed that yoga led to small or moderate improvements in low back-related functions at three and six months, compared with non-exercise controls in chronic nonspecific low back pain. However, while there are only subjective measurements in the literature about which one is more effective, there is no evidence that includes objective measurements. For this purpose, in this study, the investigators aim to determine which of the different exercises recommended for low back pain contract the muscle more effectively and compare these measurements with anthropometric measurements.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who agreed to participate in the study
* Individuals between the ages of 18-30

Exclusion Criteria:

* Individuals with congenital lumbar pathology,
* who had previously operated on the back, lumbar region
* who had scoliosis
* who had a length difference in the lower extremities

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: Individuals who agreed to participate in the study were determined as individuals between the ages of 18-30.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-03-22 (Estimated); Primary Completion 2023-04-22 (Estimated); Study Completion 2023-05-20 (Estimated)

PRIMARY OUTCOMES:
Surface EMG activations | 4 weeks
  The investigators will try to find out which of the exercises such as pressing the back back, waist extension on the balance ball, lumbar extension in the active prone position, Superman exercises have better lumbar extensor muscle activations. Muscle activations of individuals will be evaluated using superficial EMG. An 8-channel EMG Noraxon MiniDTS system (Noraxon, USA, Inc, Scottsdale, AZ) will be used to measure signals from the muscles.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided